CLINICAL TRIAL: NCT02078089
Title: A Phase Ib Study of Oxcarbazepine Plus Morphine in Patients With Refractory Cancer Pain
Brief Title: Oxcarbazepine Plus Morphine in Patients With Refractory Cancer Pain
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: Costantine Albany (Other)
Responsible Party: Sponsor-Investigator, Costantine Albany, Assistant Professor of Medicine, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IUCRO-0453
Record Dates: First submitted 2014-02-24; First posted 2014-03-05 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Cancer
Keywords: Refractory cancer pain
MeSH Terms: conditions — Neoplasms; Cancer Pain | interventions — Morphine; Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oxcarbazepine and Morphine (Other): Patients must be on stable or increasing doses of greater than or equal to 180 mg of morphine sulfate per day. Morphine is taken orally for 42 days.
  In addition to Morphine, patients will also receive oral Oxcarbazepine 150 mg, every 12 hours, for 2 weeks, then increase the dose to 300 mg, every 12 hours, for 2 weeks and then increase the dose to 450 mg, every 12 hours, for the final 2 weeks. Patients will take oral tablets of oxcarbazepine for a total of 42 days.
  Interventions: Drug: Morphine; Drug: Oxcarbazepine

INTERVENTIONS:
Drug: Morphine — Morphine will be given to patients as part of their standard care
  Other Names: Morphine Sulfate
Drug: Oxcarbazepine — Can be taken with or without food at the same time as morphine. Morphine will be provided to patients free of charge.
  Other Names: Tileptal

SUMMARY:
This is an open-label, single arm, Phase Ib dose escalation study of Oxcarbazepine with morphine in patients with refractory cancer pain. The primary endpoint is to evaluate the safety and toxicity of the combination of Oxcarbazepine plus morphine. The secondary endpoints are improving pain control, reduce morphine use and improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information.

  •≥ 18 years old at the time of informed consent
* Patients with histologically confirmed diagnosis of cancer NOTE: Patients with active cancer or post treatment are allowed on the study.
* Patients must be receiving stable or increasing doses of morphine for 1-2 weeks prior to registration for protocol therapy.

NOTE: Switching patient from current pain regimen to morphine equivalent for at least 1-2 weeks prior to registration for protocol therapy is required.

* Requiring greater than or equal to 180 mg of morphine per day. See Appendix 1 for Morphine Conversion Calculator.
* Inadequately controlled pain even with the use of morphine (VAS score >5) See Appendix 8
* Rescue pain medications are allowed this may include the use of NSAIDS or Tylenol as well as morphine IR.
* ECOG Performance Status of 0-2
* Ability to swallow and tolerate oral tablets.
* Patients getting radiation therapy are allowed at the discretion of the treating physician.
* Females of childbearing potential must have a negative pregnancy test NOTE: Females are considered of child bearing potential unless they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal (> 12 months since last menses).

NOTE: Females using hormonal contraceptives should be switched to non-hormonal forms of contraception.

The following laboratory values must be obtained. Patient with aplastic anemia will be excluded.

* White blood cell count (WBC) ≥ 3.0 K/mm3
* Absolute neutrophil count ≥ 1.5 K/mm3
* Hemoglobin (Hgb) ≥ 9 g/dL
* Platelets ≥ 75 K/mm3
* Creatinine ≤ 1.5 mg/dl
* Bilirubin ≤ 1.5 x ULN
* Aspartate aminotransferase (AST, SGOT) ≤ 3 x ULN
* Alanine aminotransferase (ALT, SGPT) ≤ 3 x ULN

Exclusion Criteria:

• Active central nervous system (CNS) metastases. Patients with neurological symptoms should undergo a head CT scan or brain MRI to exclude brain metastasis, at the discretion of the treating physician.

NOTE: Patients with prior brain metastasis may be considered if they have completed their treatment for brain metastasis, no longer require corticosteroids, and are asymptomatic.

• Concurrent use of adjuvant medication such as but not limited to: gabapentin, pregabalin or duloxetine etc.

NOTE: Patients on gabapentin or pregabalin can be considered if they can be tapered off before enrolling on the study.

* Treatment with any investigational agent within 30 days prior to registration for protocol therapy.
* Patient with rapidly escalating pain that require hospitalization or an intravenous opioid therapy
* Concurrent participation in a clinical trial which involves another investigational agent.
* Concurrent use of medications that are strong CYP3A4 inhibitors within 14 days prior to registration for protocol therapy as Oxcarbazepine is strong CYP3A4 inducer. See Appendix 7.

NOTE: Concurrent use of other CYP3A4 inhibitors may be allowed at the discretion of the treating physician or principal investigator.

* Allergic reaction to carbamazepine or oxcarbazepine (HLA-B1502)
* Allergy or other contraindication to morphine sulphate
* Opiate-induced uncontrolled constipation or bowel obstruction
* Patient who lives alone.
* Female who is pregnant or breastfeeding
* Patient who has a diagnosis of epilepsy and/or is currently taking anti-epileptic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2014-12-11 (Actual); Study Completion 2014-12-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety and toxicity | 1 year
  Evaluate the safety and toxicity of oxcarbazepine in combination with morphine

SECONDARY OUTCOMES:
Changes in Pain control | 1 year
  Evaluate changes in pain control after adding oxcarbazepine to morphine
Changes in Consumption | 1 year
  Evaluate changes morphine consumption after adding oxcarbazepine to morphine
Changes in Quality of Life | 1 year
  Evaluate changes in Quality of Life after adding oxcarbazepine to morphine

CONTACTS AND LOCATIONS:
Overall Officials: Costantine Albany, M.D., Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Indiana Univeristy Health Hospital, Indianapolis, Indiana
  - Indiana University Simon Cancer Center, Indianapolis, Indiana